CLINICAL TRIAL: NCT04433520
Title: Amplatzer™Trevisio™Delivery System Post-Approval Study
Brief Title: Trevisio Post-Approval Study
Acronym: TrevisioPAS
Status: Active, not recruiting | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: ABT-CIP_10319
Record Dates: First submitted 2020-06-12; First posted 2020-06-16 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: PFO - Patent Foramen Ovale; ASD - Atrial Septal Defect; VSD - Muscular Ventricular Septal Defect; PIVSD - Post Infarct Muscular Ventricular Septal Defect
Keywords: ABT-CIP_10319; Amplatzer Trevisio Intravascular Delivery System; Amplatzer Occluder devices
MeSH Terms: conditions — Foramen Ovale, Patent; Heart Septal Defects, Atrial

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- ASD/PFO cohort: Subjects indicated for atrial septal defect (ASD) closure with either the ASO or ASD-MF devices as well as subjects indicated for patent foramen ovale (PFO) closure with the Amplatzer PFO Occluder.
  The Amplatzer Trevisio Delivery System is to be used for facilitating percutaneous, transcatheter implantation of the occluders.
  Interventions: Device: Amplatzer™ Trevisio™ Intravascular Delivery System using Amplatzer PFO Occluder, ASO or Amplatzer Cribriform Occluder
- VSD cohort: Subjects indicated for ventricular septal defect (VSD) closure with either the MuscVSD or PIVSD occluders.
  Interventions: Device: Amplatzer™ Trevisio™ Intravascular Delivery System using Amplatzer Muscular VSD Occluder or Amplatzer Post-Infarct Muscular VSD Occluder

INTERVENTIONS:
Device: Amplatzer™ Trevisio™ Intravascular Delivery System using Amplatzer PFO Occluder, ASO or Amplatzer Cribriform Occluder — Amplatzer Trevisio Delivery System is used for facilitating percutaneous, transcatheter implantation of the Amplatzer PFO Occluder, ASO or Amplatzer Cribriform Occluder.
  Groups: ASD/PFO cohort
Device: Amplatzer™ Trevisio™ Intravascular Delivery System using Amplatzer Muscular VSD Occluder or Amplatzer Post-Infarct Muscular VSD Occluder — Amplatzer Trevisio Delivery System is used for facilitating percutaneous, transcatheter implantation of the Amplatzer Muscular VSD Occluder or Amplatzer Post-Infarct Muscular VSD Occluder.
  Groups: VSD cohort

SUMMARY:
A single-arm, non-randomized, multi-center clinical study of the Amplatzer™ Trevisio™ Intravascular Delivery System for facilitating percutaneous, transcatheter implantation of the Amplatzer™ Occluder Devices.

ELIGIBILITY:
Inclusion Criteria

1. Patient is indicated for implantation with the Amplatzer Septal Occluder for occlusion of a secundum atrial septal defect (Note: This does not include the indication for closure of a fenestration following a fenestrated Fontan procedure) OR subject is indicated for implantation with the Amplatzer PFO Occluder OR subject is indicated for implantation with the Amplatzer Muscular VSD Occluder OR subject is indicated for implantation with the Amplatzer Post-Infarct Muscular VSD Occluder
2. Patient is of legal age and has provided his/her own written, informed consent.

OR

Patient is a minor and has provided verbal and/or written informed consent or assent per local EC requirements, and his/her legally authorized representative, or representatives, have provided written informed consent on behalf of the minor according to local EC requirements

Exclusion Criteria

1. Presence of anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the Principal Investigator's opinion, could limit the subject's ability to participate in the clinical study or to comply with follow-up requirements.
2. Exclusion Criteria for Patients Undergoing ASD Closure with the Amplatzer ASO or Amplatzer ASD-MF Occluder

   * Patients known to have extensive congenital cardiac anomaly that can only be adequately repaired by cardiac surgery
   * Patients known to have sepsis within 1 month prior to implantation, or any systemic infection that cannot be successfully treated prior to device placement
   * Patients known to have demonstrated intracardiac thrombus on echocardiography (especially left atrial or left atrial appendage thrombi)
   * Patients whose size or condition (e.g., too small for transesophageal echocardiography [TEE] probe, catheter size, vasculature size, active infection) would cause the patient to be a poor candidate for cardiac catheterization
   * Patients with defect margins less than 5 mm to the coronary sinus, inferior vena cava rim, an atrioventricular valve, or the right upper lobe pulmonary vein
3. Exclusion Criteria for Patients Undergoing PFO Closure

   * Presence of thrombus at the intended site of implant, or documented evidence of venous thrombus in the vessels through which access to the defect is gained. Thrombus must be ruled out prior to introducing the delivery system.
   * Active endocarditis or other infections producing bacteremia
   * Patients whose vasculature, through which access to the defect is gained, is inadequate to accommodate the appropriate sheath size
   * Anatomy in which the Amplatzer™ PFO device size required would interfere with other intra-cardiac or intravascular structures, such as valves or pulmonary veins
   * Patients with known hypercoagulable states
   * Patients with intra-cardiac mass or vegetation, thrombus, or tumor
4. Exclusion Criteria for Patients Undergoing VSD Closure with the Amplatzer Muscular VSD Occluder or Amplatzer Post-Infarct Muscular VSD Occluder

   * Body weight <8 kg
   * Tetralogy of Fallot
   * Intracardiac thrombi on echocardiography

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This clinical study will enroll male and female adults and children with a PFO (adults only), ASD or VSD who are indicated for transcatheter closure. Patients must meet all general eligibility criteria and provide written informed consent prior to sites conducting any study-specific procedures not considered standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 251 (Estimated)
Dates: Start 2020-09-14 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Effectiveness Endpoint: Technical Success -successful deployment and release of at least one device | 5years
Safety Endpoint : Device- or procedure-related serious adverse events through discharge or 7 days, whichever occurs first | 5years
  Includes:
  * Cardiac perforation
  * Sustained atrial fibrillation requiring intervention
  * Device thrombus
  * Device erosion
  * Device embolization
  * Vascular complication requiring surgical intervention
  * Device- or procedure related serious adverse event leading to death

OTHER OUTCOMES:
Descriptive Endpoints | 5years
  * The number of times the device is recaptured
  * The number of times the device is repositioned
  * Total fluoroscopy time
  * Ease of use - investigators will be asked survey questions about their first experience with the Amplatzer Trevisio Delivery System.

CONTACTS AND LOCATIONS:
Overall Officials: Barathi Sethuraman, Study Director — DVP Global Clinical Affairs Structural Heart
Locations (22):
- France (7):
  - CHU Trousseau, Chambray-lès-Tours
  - CHU Gabriel Montpied, Clermont-Ferrand
  - Centre Médico Chirurgical Marie Lannelongue, Le Plessis-Robinson
  - CHRU Lille, Lille
  - Hopital d'adulte de la Timone, Marseille
  - CHU Hopital G. & R. Laënnec, Nantes
  - Hopital Haut Leveque, Pessac
- Germany (4):
  - Herz- und Diabeteszentrum NRW, Bad Oeynhausen
  - Deutsches Herzzentrum Berlin, Berlin
  - Universitätsklinikum Schleswig-Holstein Campus Kiel, Kiel
  - Deutsches Herzzentrum München des Freistaates Bayern, München
- Italy (3):
  - Fondazione Toscana Gabriele Monasterio Via Aurelia Sud, Massa, Tuscany
  - Azienda Ospedaliera Monaldi, Napoli
  - Policlinico San Donato, San Donato Milanese
- Amsterdam Academic Medical Centre (AMC), Amsterdam, Netherlands
- Poland (3):
  - Gornoslaskie Centrum Medyczne im.prof. Leszka Gieca ul., Katowice, Silesian Voivodeship
  - Uniwersytekie Centrum Kliniczne, Gdansk
  - The Cardinal Stefan Wyszynski Institute of Cardiology, Warsaw
- Spain (3):
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario de la Paz - Pediatrico, Madrid
  - Hospital Universitario de la Paz, Madrid
- Stadtspital Triemli, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No